CLINICAL TRIAL: NCT07343128
Title: Ultrasound-Guided Stellate Ganglion Block in Fibromyalgia: A Randomized, Single-Center, Single-Blind, Sham-Controlled Trial
Brief Title: Ultrasound-Guided Stellate Ganglion Block in Fibromyalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Yağmur Can DADAKÇI, Principal Investigator, Sanliurfa Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRU-25-1-30
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Lidocaine; Dexamethasone; dexamethasone 21-phosphate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants were randomized 1:1 to receive either ultrasound-guided SGB or a sham control procedure.
Who Masked: Participant
Masking Description: "Single-blind. Participants were blinded to treatment assignment. The investigator performing the procedures and the outcome assessors were aware of the group allocation."
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block (Experimental): Participants in this group received two ultrasound-guided stellate ganglion blocks at the C7 level, performed one week apart. Under real-time ultrasound guidance, a 22-gauge spinal needle was advanced to the stellate ganglion region. Following negative aspiration, a 7 mL mixture containing 8 mg of non-particulate dexamethasone and 2 mL of 2% lidocaine (diluted with normal saline) was injected. Success was clinically confirmed by the development of ipsilateral Horner syndrome.
  Interventions: Drug: Lidocaine and Dexamethasone
- Sham Control (Sham Comparator): Participants in this group underwent the same preparation, positioning, and ultrasound imaging as the intervention group to maintain blinding. They received two sham procedures, performed one week apart. In each procedure, 2 mL of normal saline was injected intramuscularly into the sternocleidomastoid muscle in a region distant from the stellate ganglion. This procedure replicated the needle insertion and ultrasound application without affecting the sympathetic nerves.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Lidocaine and Dexamethasone — A mixture of 2 mL of 2% lidocaine and 8 mg of non-particulate dexamethasone, diluted with normal saline to a total volume of 7 mL. Administered via ultrasound-guided injection at the C7 level. Two doses in total, with a one-week interval.
  Other Names: Lidocaine Hydrochloride, Dexamethasone Sodium Phosphate
  Arms: Stellate Ganglion Block
Other: Normal Saline — 2 mL of 0.9% normal saline administered via intramuscular injection into the sternocleidomastoid muscle. Two doses in total, with a one-week interval.
  Other Names: 0.9% Sodium Chloride, Placebo
  Arms: Sham Control

SUMMARY:
This study evaluates the efficacy and safety of ultrasound-guided stellate ganglion block (SGB) as an adjunctive treatment for patients with treatment-resistant fibromyalgia. Patients who continue to experience significant symptoms despite stable duloxetine therapy (60 mg/day) were randomized to receive either ultrasound-guided SGB or a sham control procedure. The study aims to determine if SGB can provide clinically meaningful improvements in fibromyalgia impact and pain intensity compared to a sham injection.

DETAILED DESCRIPTION:
This is a single-center, randomized, single-blind, sham-controlled trial conducted at Sanliurfa Education and Research Hospital.

Participants: Adults aged 18-65 years diagnosed with fibromyalgia (2016 ACR criteria) who have been receiving a stable dose of duloxetine 60 mg/day for at least 4 weeks but remain symptomatic.

Procedures: Participants were randomized 1:1 to either the SGB group or the sham control group.

SGB Group: Received ultrasound-guided stellate ganglion block at the C7 level using a mixture of 8 mg dexamethasone and 2 mL of 2% lidocaine (diluted to 7 mL with saline).

Sham Group: Received an intramuscular injection of 2 mL normal saline into the sternocleidomastoid muscle under ultrasound guidance.

Both groups received two procedures, performed one week apart. All patients continued their fixed-dose duloxetine throughout the study.

Assessments: The primary outcome is the change in the FIQR total score from baseline to 1 week. Secondary outcomes include FIQR changes at 1 month, pain intensity (NRS), and responder rates. This is a single-blind study where only the participants were blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia Syndrome (FMS) according to the 2016 American College of Rheumatology criteria.
* Followed for at least 1 year with insufficient benefit from previous pharmacological and/or non-pharmacological treatments.
* Receiving a stable dose of duloxetine 60 mg once daily for at least 4 weeks prior to inclusion.
* Willingness to continue the fixed dose of duloxetine throughout the study.
* Aged between 18 and 65 years.

Exclusion Criteria:

* Non-pharmacological treatments within the previous 6 months (e.g., acupuncture, ozone therapy, cognitive behavioral therapy).
* Local infection at the injection site.
* Pregnancy or suspected pregnancy.
* Known allergy to local anesthetics.
* History of malignancy.
* Bleeding or coagulation disorders or use of oral anticoagulants.
* Uncontrolled hypertension, diabetes mellitus, asthma, chronic obstructive pulmonary disease, or heart failure.
* Psychiatric or cognitive disorders that could interfere with treatment compliance (e.g., severe psychiatric illness, dementia).
* Refusal of interventional treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire Revised (FIQR) Total Score | Baseline to 1 week after the first injection
  The FIQR is a 21-item validated instrument that assesses the overall impact of fibromyalgia on physical function, overall impact, and symptoms. Total score ranges from 0 to 100, with higher scores indicating greater disease impact. Change from baseline to 1 week is the primary endpoint.

SECONDARY OUTCOMES:
Change in FIQR Total Score at 1 Month | Baseline to 1 month
  Change in FIQR total score from baseline to 1 month (3 weeks after the second injection).
Change in Numerical Rating Scale (NRS) Pain Score | Baseline, 1 week, and 1 month
  Pain intensity over the previous week assessed using an 11-point NRS (0 = no pain, 10 = worst pain imaginable). Change from baseline to 1 week and 1 month.
FIQR Responder Rates (≥30% and ≥50% Improvement) | 1 week and 1 month
  Percentage of patients achieving at least 30% and at least 50% reduction in FIQR total score from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: yagmur Dadakci, Principal Investigator — Sanliurfa Education and Research Hospital
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Şanlıurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly shared to protect participant privacy. De-identified data may be made available from the corresponding author upon reasonable request and with appropriate institutional approvals.